CLINICAL TRIAL: NCT02538718
Title: Efficacy and Safety of MgSO4 as Tocolytics Compared to Ritodrine in Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MgSO4 study
Record Dates: First submitted 2015-08-28; First posted 2015-09-02 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

ARMS (2):
- YTP(ritodrine) arm (Active Comparator): who randomly assigned to have Yutopar(ritodrine) as tocolytics
  Interventions: Drug: YTP(Ritodrine)
- MgSO4 arm (Experimental): who were randomised to have MgSO4 as tocolytics
  Interventions: Drug: MgSO4

INTERVENTIONS:
Drug: MgSO4
  Arms: MgSO4 arm
Drug: YTP(Ritodrine)
  Arms: YTP(ritodrine) arm

SUMMARY:
Ritodrine is the conventional and the only approved tocolytics in Korea(by KFDA), although it was withdrawn from the US market more than 10 years ago. As already known well, ritodrine has many side effects such as tachycardia, hyperglycemia, pulmonary edema and so on. When such complications of ritodrine appears, clinicians consider of using MgSO4 as substitute, but its use is off-the-label yet in Korea. Facing this discrepancy, the investigators want to compare the efficacy and safety of MgSO4 with ritodrine and prove that MgSO4 is not inferior to ritodrine as tocolytics. For the singleton and twin pregnancies between 24+0weeks and 34 completed weeks whose uterine contraction is more than 4 during 20 minutes period with their cervical ripening is more than 25%, the investigators randomise them in Ritodrine group or MgSO4 group. Then, the investigators will check the change of their interval of uterine contraction, degree of pain and the appearance of any side effects or treatment failure sign.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 24+0 to 34+6weeks
* singleton and twin pregnancies
* preterm labor with more than 4 times of uterine contraction for 20 minutes or more than 8 times for 1 hour on external tocography
* cervical dilatation of 0 to 3cm and cervical ripening more than 25%, or cervical length in sonography below 2cm

Exclusion Criteria:

* triplet etc
* preterm premature rupture of membrane
* cervical dilatation more than 3cm
* history of cerclage operation during this pregnancy
* placenta previa
* severe hypertensive diseases in pregnancy
* history of administration of any tocolytics 12 hours before enrollment
* fever more than 38.0'c

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
Efficacy of MgSO4 as tocolytics : increased interval of uterine contraction, decreased maternal painful sensation, stopping the cervical change | 48 hours later

CONTACTS AND LOCATIONS:
Overall Officials: Joong Shin Park, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Goverment Seoul National University Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046